CLINICAL TRIAL: NCT02979899
Title: A Randomized Phase 3 Trial of TRC105 and Pazopanib Versus Pazopanib Alone in Patients With Advanced Angiosarcoma (TAPPAS)
Brief Title: Trial of TRC105 and Pazopanib Versus Pazopanib Alone in Patients With Advanced Angiosarcoma
Acronym: TAPPAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105SAR301
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Advanced Angiosarcoma
Keywords: angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — carotuximab; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRC105 plus votrient (Experimental): weekly TRC105 i.v. in combination with standard dose votrient by mouth, once daily
  Interventions: Biological: TRC105; Drug: Votrient
- votrient (Active Comparator): standard dose votrient by mouth, once daily
  Interventions: Drug: Votrient

INTERVENTIONS:
Biological: TRC105 — TRC105 antibody
  Other Names: anti-endoglin antibody; carotuximab
  Arms: TRC105 plus votrient
Drug: Votrient — pazopanib
  Other Names: pazopanib

SUMMARY:
This is a study of TRC105 in combination with standard dose pazopanib compared to single agent pazopanib in patients with angiosarcoma not amenable to curative intent surgery (e.g., metastatic or bulky disease, and disease for which surgical resection would carry an unacceptable risk to the patient) who have not received pazopanib or TRC105 previously.

DETAILED DESCRIPTION:
TRC105 (carotuximab) is a monoclonal antibody to endoglin (CD105), an essential angiogenic target highly expressed on tumor vessels that is distinct from VEGFR. Endoglin is also expressed directly on tumor cells in angiosarcoma and is upregulated following VEGF inhibition. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models and complements the activity of bevacizumab and multi-kinase inhibitors that target the VEGFR.

Pazopanib is an oral inhibitor of multiple receptor tyrosine kinases, including vascular endothelial growth factor receptor (VEGFR)-1, VEGFR-2, and VEGFR-3 at therapeutic plasma concentrations. These receptors are implicated in pathologic angiogenesis, tumor growth, and cancer progression.

By targeting a non-VEGF pathway that is upregulated following VEGF inhibition, TRC105 has the potential to complement VEGFR tyrosine kinase inhibitors (TKIs) and could represent a major advance in the treatment of angiosarcoma. Together, the use of TRC105 with pazopanib may result in more effective angiogenesis inhibition and improved clinical efficacy over that seen with pazopanib alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed angiosarcoma that is not amenable to curative intent surgery (e.g., metastatic or bulky disease and disease for which surgical resection would carry an unacceptable risk to the patient). Pathology report will be reviewed by sponsor prior to randomization.
2. Documented progression on or following most recent systemic chemotherapy regimen (not required for chemotherapy-naïve patients), within 4 months prior to screening
3. Measurable disease by RECIST v1.1
4. Age of 18 years or older; in addition, patients age 12 to 17 years may enroll beginning in Cohort 2 if weight ≥ 40 kg
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Resolution of all acute AEs resulting from prior cancer therapies to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) grade ≤ 1 or to that patient's pre-study baseline (except alopecia or neuropathy)
7. Adequate organ function
8. Willingness and ability to consent (and assent if under age 18) for self to participate in study
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
10. Angiosarcoma tumor specimen, if available
11. Men who are sterile (including vasectomy confirmed by post vasectomy semen analysis) OR agree to use a condom with spermicide (refer to Section 2.6.1.3) and to not donate sperm during the study and for at least 180 days following last dose of TRC105 or pazopanib
12. Woman of non-child bearing potential due to surgical sterilization (at least 6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history or menopause (i.e., no menstrual bleeding for more than 12 months in a women aged 45 years or more), OR woman of child bearing potential who test negative for pregnancy at time of enrollment based on serum pregnancy test and agree to use at least 2 acceptable methods of birth control, one of which must be highly effective, during the study and for at least 180 days after stopping TRC105 or pazopanib

Exclusion Criteria:

1. Prior treatment with TRC105
2. Prior treatment with any VEGF inhibitor
3. More than two prior lines (may be combination regimens) of chemotherapy for angiosarcoma (neoadjuvant/adjuvant treatment does not count as a line of treatment)
4. Current treatment or participation on another therapeutic clinical trial
5. Women who are pregnant or breastfeeding
6. Receipt of systemic anticancer therapy, including investigational agents, within 5 times the agent's elimination half-life of starting study treatment
7. Major surgical procedure or significant traumatic injury within 4 weeks prior to randomization and must have fully recovered from any such procedure or injury; planned surgery (if applicable) or the anticipated need for a major surgical procedure within the next six months. Note: the following are not considered to be major procedures and are permitted up to 7 days before randomization: Thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, and imaging-guided biopsy for diagnostic purposes
8. Patients who have received wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvic bones or equivalent) or limited field radiation for palliation < 14 days prior to randomization
9. Uncontrolled hypertension defined as systolic > 150 or diastolic > 100 mm Hg on the average of the 3 most recent BP readings. Anti-hypertensives may be started prior to randomization.
10. Ascites or pleural effusion requiring intervention or that required intervention or recurred within three months prior to randomization
11. Pericardial effusion (except trace effusion identified by echocardiogram) within three months prior to randomization
12. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 28 days prior to randomization
13. Angina, myocardial infarction, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism , pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) within 6 months prior to randomization. Deep venous thrombosis within 3 months prior to randomization unrelated to a central venous catheter, unless the patient is anti-coagulated without the use of warfarin for at least 2 weeks prior to randomization. In this situation, low molecular weight heparin is preferred
14. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g., hereditary hemorrhagic telangiectasia). Patients with bleeding cutaneous lesions not actively requiring transfusions are eligible. Patients who have been uneventfully anti-coagulated with low molecular weight heparin are eligible
15. Hemoptysis (> ½ teaspoon [2.5 mL] of bright red blood) within 6 months prior to randomization
16. Thrombolytic use (except to maintain i.v. catheters) within 10 days prior to randomization
17. Known active viral or nonviral hepatitis or cirrhosis
18. Peptic ulcer within the past 3 months prior to randomization, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD)
19. Presence of tumor(s) invading into the heart or great vessels (including carotid artery) or another location where bleeding is associated with high morbidity including patients with primary cardiac or great vessel angiosarcoma
20. Gastrointestinal perforation or fistula in the 6 months prior to randomization unless underlying risk has been resolved (e.g., through surgical resection or repair)
21. Presence of a malabsorption syndrome, gastrointestinal disorder, or gastrointestinal surgery that could affect the absorption of pazopanib
22. History of prior malignancy except adequately treated basal cell or squamous cell skin cancer or adequately treated, with curative intent, cancer from which the patient is currently in complete remission per Investigator's judgment; patients with history of breast cancer and no evidence of disease on hormonal therapy to prevent recurrence and patients with prostate cancer on adjuvant hormonal therapy with undetectable PSA are eligible
23. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
24. Active infection that requires systemic treatment
25. Concurrent use or receipt of a strong CYP3A4 inducer within 12 days prior to randomization or a strong CYP3A4 inhibitor within 7 days prior to randomization (see Table 10)
26. History of severe hypersensitivity reaction to any monoclonal antibody
27. Other severe acute or chronic medical (including bone marrow suppressive diseases) or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, impede the ability of the patient to complete all protocol-specified activities, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, Study Director — TRACON Pharmaceuticals
Locations (39):
- United States (26):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Sandy Springs, Georgia
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health, Lake Success, New York
  - MSKCC, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washinton, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Medical University,Vienna, Vienna, Austria
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Helios Klinikum, Bad Saarow
  - Mannheim University Medical Center, Mannheim
  - Klinikum derUniversitat Munchen, Munich
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Spain (2):
  - Institut Català d'Oncologia (ICO), Barcelona
  - 12 de Octubre University Hospital, Madrid
- Royal Marsden NHS, Chelsea, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones RL, Ravi V, Brohl AS, Chawla S, Ganjoo KN, Italiano A, Attia S, Burgess MA, Thornton K, Cranmer LD, Cheang MCU, Liu L, Robertson L, Adams B, Theuer C, Maki RG. Efficacy and Safety of TRC105 Plus Pazopanib vs Pazopanib Alone for Treatment of Patients With Advanced Angiosarcoma: A Randomized Clinical Trial. JAMA Oncol. 2022 May 1;8(5):740-747. doi: 10.1001/jamaoncol.2021.3547. PMID 35357396
- [Derived] Mehta CR, Liu L, Theuer C. An adaptive population enrichment phase III trial of TRC105 and pazopanib versus pazopanib alone in patients with advanced angiosarcoma (TAPPAS trial). Ann Oncol. 2019 Jan 1;30(1):103-108. doi: 10.1093/annonc/mdy464. PMID 30357394

RESULTS

PARTICIPANT FLOW:
Groups:
- TRC105 + Votrient: Weekly TRC105 i.v. in combination with standard dose votrient by mouth, once daily
  TRC105: TRC105 antibody
  Votrient: pazopanib
Period: Overall Study
Arm/Group | TRC105 + Votrient | Votrient
Started | 64 | 64
Completed | 64 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRC105 + Votrient | Votrient | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Median (Full Range); unit: years] | 69 [32 to 82] | 67 [25 to 84] | 68 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 42 | 77
  Male | 29 | 22 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 55 | 56 | 111
  Not Reported | 1 | 1 | 2
  Unknown | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 50 | 46 | 96
  Poland | 0 | 4 | 4
  United Kingdom | 8 | 9 | 17
  France | 6 | 5 | 11
ECOG Performance Status [Count of Participants; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. = Dead
  Participants
    ECOG Grade 0 | 30 | 27 | 57
    ECOG Grade 1 | 32 | 36 | 68
    Not Available | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival of Patients With Unresectable Angiosarcoma
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Progression free survival is defined as time from randomization to either first disease progression (per independent radiology review of images by RECIST 1.1) or death from any cause.
Time Frame: from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to cut off date of interim analysis (25 months)
Population: All patients randomized onto study by cut off date of interim analysis
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | TRC105 + Votrient | Votrient
Number analyzed (Participants) | 62 | 61
months
  PFS by RECIST 1.1 | 4.2 [2.8 to 8.3] | 4.3 [2.9 to NA] — Confidence interval not estimable because not enough events to estimate a standard error
  PFS by Investigator Assessment | 3.5 [2.6 to 5.5] | 2.9 [2.6 to 4.1]

2. Secondary Outcome: Objective Response Rate of Patients With Unresectable Angiosarcoma
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR) is disappearance of all target lesions; Partial Response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Overall response rate is defined as the number of patients with a best response designation of complete response or partial response recorded between the date of randomization and the date of documented progression.
Time Frame: as for outcome 1
Population: All patients randomized onto study by cut off date of interim analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 + Votrient | Votrient
Number analyzed (Participants) | 62 | 61
Participants | 3 | 8

3. Secondary Outcome: Overall Survival of Patients With Unresectable Angiosarcoma
Description: Overall survival is the number of death events at 25 months, including all on-study and off-study deaths (past post-treatment 28-day follow up visit)
Time Frame: from beginning of study to cut off date of interim analysis (25 months)
Population: All patients randomized onto study by cut off date of interim analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 + Votrient | Votrient
Number analyzed (Participants) | 62 | 61
Participants | 17 | 19

4. Secondary Outcome: To Characterize Patient Reported Outcomes Between the Two Arms of the Study
Description: Patient reported outcomes as measured by the EuroQol five dimensions questionnaire (EQ-5D-5L) and the European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30). The EORTC QLQ-C30 health scale is on a scale of 1 to 7, with 1 being poor health and 7 being excellent health. The EQ-5D-5L scale is on a scale of 0 to 100, with 0 being the worst health one can imagine, and 100 being the best health one can imagine.
Time Frame: Screening and 9 weeks (Cycle 3 Day 1)
Population: All patients who completed the questionnaire during specified intervals listed below
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TRC105 + Votrient | Votrient
Number analyzed (Participants) | 64 | 62
units on a scale
  EORTC QLQ-C30 Health Score at Screening | 5 [1 to 7] | 5 [1 to 7]
  EQ-5D-5L Health Score at Screening: number analyzed (Participants) | 59 | 54
  EQ-5D-5L Health Score at Screening | 75 [5 to 100] | 75 [20 to 100]
  EORTC QLQ-C30 Health Score at Cycle 3 Day 1: number analyzed (Participants) | 39 | 38
  EORTC QLQ-C30 Health Score at Cycle 3 Day 1 | 4 [1 to 6] | 5 [1 to 6]
  EQ-5D-5L Health Score at Cycle 3 Day 1: number analyzed (Participants) | 38 | 38
  EQ-5D-5L Health Score at Cycle 3 Day 1 | 70 [20 to 100] | 70 [20 to 97]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire duration of the study (a period of 26 months).
Description: AEs were collected for each patient that received at least 1 dose of study drug from informed consent through 28 days following the last dose of study drug. Related AEs were followed until they resolved or became stable. All-Cause Mortality was monitored in all randomized participants as overall survival (OS) was a secondary endpoint of the study. OS was followed until death regardless of subsequent treatment. Patients were eligible for participation in the trial until they progressed.
Groups:
- TRC105 + Votrient: All patients that received at least one dose of TRC105 in combination with pazopanib
- Votrient: All patients that received at least one dose of pazopanib alone.
Arm/Group | TRC105 + Votrient | Votrient
All-Cause Mortality (participants affected / at risk) | 23/64 | 20/64
Serious Adverse Events (participants affected / at risk) | 27/63 | 12/57
Other Adverse Events (participants affected / at risk) | 63/63 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRC105 + Votrient (N=63) | Votrient (N=57)
Disease Progression (General disorders) | 4 | 0
Embolism (Vascular disorders) | 3 | 0
Wound infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 3
Fatigue (General disorders) | 3 | 0
Pyrexia (Gastrointestinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mental Status Change (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Tumor Hemorrhage (Nervous system disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Meningitis Aseptic (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Hematemesis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Platelet Disorder (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRC105 + Votrient (N=63) | Votrient (N=57)
Fatigue (General disorders) | 42 | 33
Diarrhea (Gastrointestinal disorders) | 38 | 31
Nausea (Gastrointestinal disorders) | 34 | 26
Hypertension (Vascular disorders) | 24 | 32
Headache (Nervous system disorders) | 42 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 26 | 19
Vomiting (Gastrointestinal disorders) | 25 | 13
Anemia (Blood and lymphatic system disorders) | 33 | 5
Weight Decreased (Investigations) | 23 | 10
Dysgeusia (Nervous system disorders) | 15 | 15
Aspartate Aminotransferase Increased (Investigations) | 16 | 14
Alanine Aminotransferase Increased (Investigations) | 15 | 12
Abdominal Pain (Gastrointestinal disorders) | 14 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Constipation (Gastrointestinal disorders) | 13 | 9
Stomatitis (Gastrointestinal disorders) | 16 | 5
Gingival Bleeding (Gastrointestinal disorders) | 17 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 6
Edema Peripheral (General disorders) | 13 | 6
Hypokalemia (Metabolism and nutrition disorders) | 14 | 4
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 9 | 9
Hypothyroidism (Endocrine disorders) | 11 | 5
Platelet Count Decreased (Investigations) | 9 | 7
Pyrexia (General disorders) | 11 | 4
Lipase Increased (Investigations) | 9 | 6
Blood Bilirubin Increased (Investigations) | 6 | 9
Hypotension (Vascular disorders) | 11 | 3
Chills (General disorders) | 10 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Dehydration (Metabolism and nutrition disorders) | 10 | 3
Flushing (Vascular disorders) | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 7 | 5
Urinary Tract Infection (Infections and infestations) | 9 | 2
Mucosal Inflammation (General disorders) | 7 | 4
Anxiety (Psychiatric disorders) | 6 | 5
Vision Blurred (Eye disorders) | 6 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 1
Insomnia (Psychiatric disorders) | 7 | 3
Dizziness (Nervous system disorders) | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 3
Blood Thyroid Stimulating Hormone Increased (Investigations) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Infusion Related Reaction (Injury, poisoning and procedural complications) | 8 | 1
Asthenia (General disorders) | 7 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 6 | 3
Dry Mouth (Gastrointestinal disorders) | 6 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Neutrophil Count Decreased (Investigations) | 5 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 6
Blood Alkaline Phosphatase Increased (Investigations) | 7 | 1
Lymphocyte Count Decreased (Investigations) | 7 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3
Fall (Injury, poisoning and procedural complications) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 5
Proteinuria (Renal and urinary disorders) | 3 | 5
Mouth Hemorrhage (Gastrointestinal disorders) | 7 | 0
Oral Pain (Gastrointestinal disorders) | 6 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 3
Blood Creatinine Increased (Investigations) | 3 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Flatulence (Gastrointestinal disorders) | 2 | 5
Embolism (Vascular disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pain (General disorders) | 5 | 1
White Blood Cell Count Decreased (Investigations) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Blood Amylase Increased (Investigations) | 3 | 3
Sinus Tachycardia (Cardiac disorders) | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
Telangiectasia (Skin and subcutaneous tissue disorders) | 5 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 0
Hypoxia (Metabolism and nutrition disorders) | 4 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Chest Pain (General disorders) | 4 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 2 | 3
Abdominal Distension (Gastrointestinal disorders) | 2 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Migraine (Nervous system disorders) | 4 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 0
Disease Progression (General disorders) | 4 | 0
Gingival Pain (Gastrointestinal disorders) | 4 | 0
Hematemesis (Gastrointestinal disorders) | 4 | 0
Lacrimation Increased (Eye disorders) | 4 | 0
Bradycardia (Cardiac disorders) | 4 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 3
Sepsis (Infections and infestations) | 0 | 3
Non-Cardiac Chest Pain (General disorders) | 3 | 2
Oral Dysesthesia (Gastrointestinal disorders) | 3 | 2
Pain Of Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Hematuria (Renal and urinary disorders) | 3 | 1
Depression (Psychiatric disorders) | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
Facial Pain (General disorders) | 3 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 1
Hyperthyroidism (Endocrine disorders) | 3 | 1
Tachycardia (Cardiac disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT02979899/Prot_SAP_000.pdf